CLINICAL TRIAL: NCT04232696
Title: Clinical Study of Neuspera's Implantable Sacral Nerve Stimulation (SNS) System in Patients With Symptoms of Urinary Urgency Incontinence (UUI)
Brief Title: Neuspera's Implantable Sacral Nerve Stimulation System in Patients With Symptoms of Urinary Urgency Incontinence (UUI)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuspera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neuspera Medical (NSM)-004; SANS-UUI (Other: Neuspera)
Record Dates: First submitted 2019-12-09; First posted 2020-01-18 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Urinary Urgency Incontinence
Keywords: UUI

STUDY DESIGN:
Intervention Model Description: Prospective, seamless two-phased pivotal study design. Phase I is designed to assess the initial feasibility of Neuspera's Implantable SNS System and to determine optimal daily stimulation parameters for Phase II. The data from Phase I informed the duration of daily stimulation and was applied in Phase II, which aims to evaluate the safety and efficacy of the system. Phase I and Phase II involve distinct patient populations with no overlap.
  Phase I enrolled 89 subjects and Phase II enrolled 242 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Neuspera Implantable Sacral Nerve Stimulation System (Experimental): Implantation of the stimulator.
  Interventions: Device: Neuspera Implantable Sacral Nerve Stimulation System

INTERVENTIONS:
Device: Neuspera Implantable Sacral Nerve Stimulation System — Stimulation of the Sacral Nerve.

SUMMARY:
Prospective, multi-center, single-arm, seamless phase-pivotal study conducted in participants diagnosed with UUI who have failed or could not tolerate more conservative treatment. The trial will be conducted in two phases.

Objective of Phase I: To assess the utilization of the system during the Sacral Nerve Stimulation (SNS) trial period and to help inform the length of hours of daily stimulation to be used in Phase II of the trial.

Objective of Phase II: To assess the safety and efficacy of the Neuspera SNS System at 6-months for the primary efficacy endpoint and at 12 months for secondary safety and efficacy endpoints.

DETAILED DESCRIPTION:
Neuspera's Implantable Sacral Nerve Stimulation (SNS) System is indicated to treat participants with UUI who have failed or could not tolerate more conservative treatments.

The study will be conducted in two phases: Phase I of the study will be conducted at up to 9 clinical study sites in the US and Europe. Phase II of the study will be conducted in up to 35 clinical sites in the US and Europe, inclusive of the Phase I centers.

Prospective, multi-center, single-arm, seamless phase-pivotal study. Objective of Phase I: To assess the utilization of the system during the Sacral Nerve Stimulation (SNS) trial period and to help inform the length of hours of daily stimulation to be used in Phase II of the trial.

Objective of Phase II: To assess the safety and efficacy of the Neuspera SNS System at 6-months for the primary efficacy endpoint and at 12 months for secondary safety and efficacy endpoints. All participants will receive the same length of device stimulation as determined in Phase I testing.

Phase I will enroll up to 55 participants. Phase II will enroll up to 255 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Has a Body Mass Index (BMI) between 18 and 40.
2. Has a diagnosis of UUI for greater than or equal to 6 months prior to the screening baseline visit date.
3. Has failed or was not a candidate for more conservative treatment (e.g. pelvic floor training, biofeedback, behavioral modification).
4. Has failed or could not tolerate (stopped taking medication due to lack of efficacy or intolerable side effects) or not a good candidate for (as determined by treating physician) at least one (1) antimuscarinic or β3 adrenoceptor agonist medication.
5. Has a diagnosis of UUI with at least 4 UUI episodes on a 72-hour diary, and minimum of one (1) UUI episode per 24-hour period.

Exclusion Criteria:

1. Has a hemoglobin A1c of greater than 8 percent, or has diabetes mellitus with glucosuria.
2. Has diabetic neuropathy.
3. Has interstitial cystitis or bladder pain syndrome as defined by either American Urological Association (AUA) or European Association of Urology (EAU) guidelines, chronic pelvic pain or recurrent symptomatic urinary tract infections.
4. Has neurogenic bladder dysfunction such as traumatic or atraumatic myelopathy, multiple sclerosis, Parkinsonism, or history of cerebrovascular accident.
5. Has documented urinary retention within 6 months prior to the screening baseline visit date.
6. Has clinically significant bladder outlet obstruction.
7. Is a subject with a mechanical obstruction such as benign prostatic hypertrophy, urethral stricture or cancer.
8. Has primary stress incontinence or mixed incontinence where the stress component predominates or has been treated surgically for stress urinary incontinence within 6 months prior to the screening baseline visit date.
9. Has received tibial nerve stimulation (TNS) in the past 3 months for the treatment of overactive bladder or unwilling to stay off TNS therapy for 12-month period following implant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Padron, MD, Principal Investigator — Florida Urology Partners
Locations (34):
- United States (31):
  - Genesis Healthcare Partners, Encinitas, California
  - Kaiser Permanente, LAMC, Los Angeles, California
  - Kaiser Permanente, San Diego, California
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Florida Urology Partners, LLC, Tampa, Florida
  - Midtown Urology, Atlanta, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Women's Health Advantage, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - UofL Health System (University of Louisville), Louisville, Kentucky
  - Ochsner Medical, New Orleans, Louisiana
  - University of Michigan Health - West, Wyoming, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Minnesota Urology, Woodbury, Minnesota
  - Specialty Research of St. Louis, St Louis, Missouri
  - Adult & Pediatric Urology P.C., Omaha, Nebraska
  - Weill Cornell Medical College, New York, New York
  - Premier Medical Group, Poughkeepsie, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - MetroHealth, Cleveland, Ohio
  - The Oregon Clinic Urogynecology West, Portland, Oregon
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, North Wales, Pennsylvania
  - Southern shores urogynecology, Myrtle Beach, South Carolina
  - Southern Urogynecology, West Columbia, South Carolina
  - Center for Pelvic Health, Franklin, Tennessee
  - Urology Austin, Austin, Texas
  - Urology Clinics of North Texas (Dallas Center for Pelvic Medicine), Dallas, Texas
  - Virginia Mason, Seattle, Washington
  - University of Washington, Seattle, Washington
- Universiteit Antwerpen, Antwerp, Belgium
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share information.

REFERENCES:
- See also: Neuspera Medical web page — http://neuspera.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ph I Study: Of 89 subjects consented, 39 subjects had implant attempted, 34 were successfully implanted. 35 subjects were screen failures, 11 withdrew consent, 1 withdrawn by investigator, 2 LTF, and 1 other withdrawal reason. Ph II Study: Of 242 subjects consented, 130 subjects had implant attempted and 128 were successfully implanted. 80 subjects were screen failure,16 withdrew consent, 3 withdrawn by investigator, 5 LTF, 4 due to site termination by sponsor, and 4 other withdrawal reasons.
Groups:
- Phase I, Neuspera Implantable Sacral Nerve Stimulation System; Phase II, Neuspera Implantable Sacral Nerve Stimulation System: Implantation of the Stimulator.
  Neuspera Implantable Sacral Nerve Stimulation System: Stimulation of the Sacral Nerve.
Period: Overall Study
Arm/Group | Phase I, Neuspera Implantable Sacral Nerve Stimulation System | Phase II, Neuspera Implantable Sacral Nerve Stimulation System
Started | 39 | 130
Completed (6 month primary endpoint timepoint) | 34 | 111
Not Completed | 5 | 19
Not completed — Implant attempted but not completed | 5 | 2
Not completed — Not satisfied with therapy outcome | 0 | 8
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Missed Visit | 0 | 2
Not completed — Other reason | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Neuspera Implantable Sacral Nerve Stimulation System; Phase II: Neuspera Implantable Sacral Nerve Stimulation System: Implantation of the simulator. Neuspera Implantable Sacral Nerve Stimulation System: Stimulation of the Sacral Nerve.
- Total: Total of all reporting groups
Arm/Group | Phase I: Neuspera Implantable Sacral Nerve Stimulation System | Phase II: Neuspera Implantable Sacral Nerve Stimulation System | Total
Number analyzed (Participants) | 39 | 130 | 169
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (12.6) | 60.4 (10.2) | 60.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 128 | 165
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 10 | 11
  Not Hispanic or Latino | 38 | 120 | 158
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 38 | 124 | 162
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30 (5.4) | 29.5 (5.1) | 29.6 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Percentage of Participants Who Experience a 50 Percent or More Change in Urinary Urgency Incontinence Episodes.
Description: Change in Urinary Urgency Incontinence episodes at six months, relative to the number of Urinary Urgency Incontinence episodes at baseline.
Time Frame: 6 months
Population: Completers data: number of subjects with completed assessments for primary endpoint
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I, Neuspera Implantable Sacral Nerve Stimulation System | Phase II, Neuspera Implantable Sacral Nerve Stimulation System
Number analyzed (Participants) | 30 | 111
percentage of participants | 93.3 [77.9 to 99.2] | 95.5 [89.8 to 98.5]

2. Primary Outcome: Primary Safety Endpoint: Defined as the Proportion of Subjects Experiencing a Device-related Serious Adverse Events.
Description: The analysis of the endpoint is the proportion of subjects experiencing a device-related SAE through the 6-month post-implant.
Time Frame: 6 months
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Neuspera Implantable Sacral Nerve Stimulation System | Phase II, Neuspera Implantable Sacral Nerve Stimulation System
Number analyzed (Participants) | 39 | 130
Participants | 0 | 0

3. Secondary Outcome: Phase II Change in Quality of Life: Measured From Baseline as Measured and Assessed by the Total and Subset International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life Score.
Description: Change from baseline in qualify of life. Total score (25 min,160 max) with higher score indicating increase impact on quality of life.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Phase II Efficacy Endpoint: Defined as the Percentage of Participants Who Experience a 50 Percent or More Change in Urinary Urgency Incontinence.
Description: Change in Urinary Urgency Incontinence episodes at 12 months post-completion of the trial phase, relative to the number of Urinary Urgency Incontinence episodes at baseline prior to the trial phase.
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Phase II Urgent Voids Per Day
Description: Change in urgent voids per day from baseline to 6-months and 12 months. Calculated across all diary episodes with at least mild urgency.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Phase II Change in Average Number of Daily Voids
Description: Change in average number of daily voids from baseline in subjects with at least 8 voids at baseline.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Phase II Comprehensive Summary of All Adverse Events
Description: The incidence of adverse events will be reported.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Phase II Device Parameter Information Collected
Description: Device amplitude will be collected in volts.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Phase II Physician and Subject User Experience Questionnaire
Description: Physician and subject satisfaction will be obtained by answering questions on the use of the device using a five point scale:strongly agree, agree, neither agree nor disagree, disagree, strongly disagree. Answers towards strongly agree indicate a better outcome.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Phase II Urinary Tract Symptoms Questionnaire: International Consultation on Incontinence Questionnaire Female & Male Lower Urinary Tract Symptoms Modules
Description: Change in female lower urinary tract symptoms questionnaire. Male questionnaire score ranges from 0-52 and female questionnaire score ranges from 0-48. Higher number indicates worse outcome.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

11. Secondary Outcome: Phase II Safety Endpoint: Defined as the Incidence of Device-related Serious Adverse Events in the Post-trial Period Follow-up.
Description: The number of serious adverse events related to the device.
Time Frame: 12 months
Reporting Status: Not Posted

12. Secondary Outcome: Phase II Urinary Output
Description: Total urinary output as measured by 72-hour bladder diary.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

13. Secondary Outcome: Phase II Fecal Incontinence Measured by Wexner Scale
Description: Wexner scale total points 0-20, higher the score the worse the outcome. Fecal incontinence as measured by the Wexner Scale compared to baseline.
Time Frame: 6 months
Reporting Status: Not Posted

14. Secondary Outcome: Phase II Patient Global Impression of Improvement
Description: Patient Global Impression of Improvement measured after implant during follow-up. Single question answered on a seven point scale: very much better, much better, a little better, no change, a little worse, much worse, very much worse. Selection of very much better is the best outcome.
Time Frame: 6 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At least 6 months post-implant
Groups:
- Ph I, Neuspera Implantable Sacral Nerve Stimulation System: Phase I, Implantation of the stimulator. Neuspera Implantable Sacral Nerve Stimulation System: Stimulation of the Sacral Nerve.
- Ph II, Neuspera Implantable Sacral Nerve Stimulation System: Implantation of the stimulator. Neuspera Implantable Sacral Nerve Stimulation System: Stimulation of the Sacral Nerve.
Arm/Group | Ph I, Neuspera Implantable Sacral Nerve Stimulation System | Ph II, Neuspera Implantable Sacral Nerve Stimulation System
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/130
Serious Adverse Events (participants affected / at risk) | 1/39 | 16/130
Other Adverse Events (participants affected / at risk) | 10/39 | 0/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I, Neuspera Implantable Sacral Nerve Stimulation System (N=39) | Ph II, Neuspera Implantable Sacral Nerve Stimulation System (N=130)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Breast Cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Post procedural stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) — Not related to Study Device or Study Procedure
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2) — Not related to Study Device or Study Procedure
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Possibly related to the implant procedure
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Shoulder Operation (Surgical and medical procedures) | 0 (0) | 1 (1) — Not related to Study Device or Study Procedure
Numbness and tingling in left foot (Nervous system disorders) | 1 (1) | 0 (0) — Not related to Study Device or Study Procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I, Neuspera Implantable Sacral Nerve Stimulation System (N=39) | Ph II, Neuspera Implantable Sacral Nerve Stimulation System (N=130)
Implant Site Pain (General disorders) | 5 (7) | NA
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Device Dislocation (Product Issues) | 3 (3) | NA
Device Breakage (Product Issues) | 2 (3) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT04232696/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT04232696/SAP_001.pdf